CLINICAL TRIAL: NCT04633200
Title: Mhealth for Pre-exposure Prophylaxis Adherence by Young Adult MSM
Brief Title: Mhealth for PrEP Adherence by Young Adult MSM, Phase 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environment and Health Group, Inc. (Industry)
Responsible Party: Principal Investigator, Patricia Weitzman, Senior Scientist, Environment and Health Group, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44MH112221-02 (NIH)
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Results first posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will receive a mobile app to support their daily PrEP adherence.
  Interventions: Other: DOT mobile app
- Control (No Intervention): Participants in the control group will receive a 2-page PrEP patient education document based information about PrEP from on the CDC website.

INTERVENTIONS:
Other: DOT mobile app — DOT is a mobile phone app that has daily pill reminders and supportive texts, as well as various features designed to support PrEP medication adherence.
  Arms: Intervention

SUMMARY:
This Phase 2 project aims to enhance and test a mobile health intervention designed to increase adherence to the daily PrEP pill among culturally-diverse young adult men who have sex with men. The intervention will include: a) personalized PrEP pill reminders b) culturally- and developmentally-sensitive text messages targeting patient education, motivation, and stress c) a gamification avatar and d) a linked online community of peers. Effectively promoting PrEP adherence would reduce new HIV infections in this at-risk population, which is subject to health disparities

DETAILED DESCRIPTION:
The project is to develop and test the effectiveness of an individually-tailored, developmentally- and culturally-sensitive, mobile health (mhealth) PrEP adherence intervention called DOT. The intervention will target culturally-diverse, young adult men, ages 18-35, who have sex with men (YMSM). The recent rise in HIV infection among young people, particularly minority YMSM, points to the value of PrEP uptake and adherence support for YMSM. In PrEP efficacy trials, younger age was the most consistent correlate with low PrEP adherence. Our DOT mhealth intervention reflects a developmental understanding of young adult decision-making, and is uniquely combined with principles from social cognitive theory, positive psychology and behavioral economics. The proposed project is based on Dr. Weitzman's successful Phase 1 trial of DOT, which led to significant improvements in PrEP adherence, PrEP treatment self-efficacy, and intention to follow PrEP treatment guidelines among the YMSM that used DOT for six weeks. Our proposed Phase 2 DOT mhealth intervention is directly responsive to Phase 1 findings by adding: 1) texts targeting motivation, patient education, and stress burden 2) online community for social support 3) linkage to the federal crisis text line 4) virtual avatar 5) cloud-based platform to view user engagement 7) calendar for clinic appointments and pharmacy refills 8) enhanced personalization of pill reminders and 9) enhanced adherence graphing. In Phase 2, we will test the effectiveness of DOT at improving PrEP adherence in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria: (self report) Individuals who self-identify as a male, age 18-35, who has sex with men or who self-identify as a bisexual male or a gay male; currently taking PrEP; own a smartphone and desirous of adherence support.

-

Exclusion Criteria: (self report) Males who do not meet the above criteria and/or currently use I.V. drugs.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 108 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Environment and Health Group, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 57 | 51
Completed | 54 | 46
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.74 (4.43) | 27.67 (4.25) | 27.17 (4.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 46 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 27
  Not Hispanic or Latino | 40 | 32 | 72
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 34 | 30 | 64
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 54 | 46 | 100

OUTCOME MEASURES:

1. Primary Outcome: Wilson Self-reported Medication Adherence Scale
Description: The self-reported medication adherence scale, developed by Wilson et al. (2016), is designed to assess self-reported medication adherence to HIV-related and other types of medications. In this study, it was used to assess self-reported PrEP medication adherence. Minimum score=0, maximum=299.9. Higher score means better adherence.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 46
score on a scale | 77.48 (13.68) | 71.59 (17.07)

2. Secondary Outcome: PrEP Medication Adherence Self Efficacy Scale
Description: This scale was adapted by Kogelman and Weitzman from the Johnson HIV Adherence Self-Efficacy Scale. The PrEP medication adherence self efficacy scale was developed to assess one's confidence in one's ability to adhere to their PrEP medication treatment plan. The minimum score = 0, maximum score =80. Higher score indicates greater PrEP medication adherence self efficacy.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 46
score on a scale | 8.26 (1.55) | 7.63 (1.82)

3. Secondary Outcome: Intention to Follow PrEP Treatment Guidelines
Description: This measure was developed by Kogelman and Weitzman to assess an individual's intention to engage in key behaviors that are recommended while on PrEP treatment, e.g. concomitant use of condoms and testing for HIV every 3 months. The minimum score=0, the maximum score=16. Higher score means greater intention to follow PrEP treatment guidelines.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 46
score on a scale | 4.26 (0.72) | 3.93 (0.95)

4. Secondary Outcome: PrEP Medication Knowledge Measure
Description: This measure was developed by Kogelman and Weitzman to assess an individual's knowledge of PrEP medication through questions about medication purpose, side effects, etc. Minimum score =0, maximum score = 8. Higher score means greater knowledge about PrEP medication.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 46
score on a scale | 6.75 (1.12) | 6.92 (1.11)

5. Secondary Outcome: Perceived Stress Scale
Description: The Perceived Stress Scale, developed by Cohen et al. (1983), is designed to measure the degree to which one perceives situations in one's life as stressful. The minimum score=0, maximum score=40. Higher score indicates higher perceived stress.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 54 | 46
score on a scale | 2.19 (0.54) | 2.28 (0.59)

ADVERSE EVENTS:
Time Frame: 12 week study period
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/51
Other Adverse Events (participants affected / at risk) | 0/57 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT04633200/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04633200/SAP_001.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04633200/ICF_002.pdf